CLINICAL TRIAL: NCT00555295
Title: Survival After Laparoscopic Colorectal Surgery
Brief Title: Laparoscopic Colorectal Surgery For Cancer- Long Term Survival
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-AS-389-CTIL
Record Dates: First submitted 2007-10-27; First posted 2007-11-08 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-06

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Colonic Resection
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the survival after laparoscopic colectomies due to carcinoma.

DETAILED DESCRIPTION:
Laparoscopic procedures for Colorectal Carcinoma are taking place in the modern era of surgery, It was not proven yet to show pure advantage over the open colectomies.

These Procedures require highly skilled stuff with long learning curve, Financial sources,Increasing operation length.

This retrospective study intends to show that the outcome of the overall survival is better in Laparoscopic patients.

All data about patients who had laparoscopic colectomies due to carcinoma in Surgery A department in Souraski Medical Center was recorded prospectively since the operation day till discharge.

The retrospective follow up will be collected from the outpatient clinic, the Oncology clinic and by questionnare to the patients.

We wish to show that patients who were operated laparoscopy have better survival, better quality of life postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of colon

Exclusion Criteria:

* Non curative operation
* Non cancerous subjects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Colon Cancer
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Avital, md, Study Chair — Tel Aviv Souraski Medical Center; Smadar Nir, md, Principal Investigator — Tel Aviv Souraski Medical Center